CLINICAL TRIAL: NCT06686134
Title: Comprehensive Clinical Evaluation Study of GLP-1RA
Status: Recruiting | Type: Observational
Sponsor: LI YAN (Other)
Responsible Party: Sponsor-Investigator, LI YAN, Chief Pharmacist, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: QFS-LY-2024-GLP-1RA-001
Record Dates: First submitted 2024-11-01; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: T2DM
Keywords: GLP1-RA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- liraglutide
- Dulagoside
- Polyethylene glycol losenatide
- Semaglutide

SUMMARY:
The objective of this project is to identify the most efficacious glucagon-like peptide-1 receptor agonists (GLP-1RAs) for the treatment of adult patients with type 2 diabetes mellitus (T2DM). In accordance with the index system and evaluation rules set forth in the Management Guidelines for Comprehensive Clinical Evaluation of Drugs, the effects of GLP-1RAs drugs in real-world settings are tracked, summarised, and analysed across six dimensions: safety, effectiveness, economy, innovation, appropriateness, and accessibility. This is done with the objective of ensuring that these drugs are fully utilised in accordance with their potential benefits. The objective is to ascertain the role of medical institutions as the principal entity responsible for the comprehensive evaluation of the clinical application of drugs and to provide data that will reduce the risk of using GLP-1RAs drugs. Moreover, the objective is to ascertain the advantages of their clinical application and to guarantee the safe and rational use of drugs for patients with type 2 diabetes mellitus. The objective of this study is to facilitate the fulfilment of medical institutions' role as the primary entity responsible for the comprehensive evaluation of the clinical application of medicines. Furthermore, the study will provide data that can be used to reduce the risk of using GLP-1RAs drugs, explore the advantages of their clinical application, and guarantee the safe and rational use of medicines for patients with type 2 diabetes.

DETAILED DESCRIPTION:
This study employed a prospective cohort design and included patients with type 2 diabetes mellitus (T2DM) who were receiving treatment with liraglutide, dulaglutide, polyethylene glycol losenatide, or simethicone. The subjects' basic information was collected, including their hospitalisation number, name, gender, age, date of birth, ethnicity, and occupation. Furthermore, data pertaining to the subjects' lifestyle habits were collected, including their history of smoking and alcohol consumption. Information pertaining to the circumstances of their hospitalisation was also collated, including the time, number, route, department, and diagnosis. Furthermore, data regarding the subjects' diabetic complications and past medical history were collected. Lastly, the time of discharge and diagnosis were recorded.

1. Collection of information on hospitalization:

   * General information: basic information (hospitalization number, name, gender, age, date of birth, ethnicity, occupation), lifestyle information (history of smoking, history of alcohol consumption), admission (admission time, number, route, department, diagnosis), information on diabetic complications and past medical history, and discharge (discharge time and diagnosis).

     ② The data presented herewith pertain to the admission test. The data set includes basic information such as height, weight, body mass index (BMI), blood pressure, and temperature. Additionally, it encompasses glucose metabolism indicators, including fasting glucose, 2-hour postprandial glucose, and glycated hemoglobin. It also includes lipid metabolism indicators, such as triglycerides and total cholesterol. Furthermore, the examination of high-density and low-density lipoproteins, electrolytes (potassium, sodium, magnesium, calcium ion concentration), and indicators of hepatic and renal function (glutamic acid aminotransferase, glutamic oxaloquatamidase) is essential. Furthermore, the following biochemical parameters were analysed: total bile acid, total bilirubin, direct bilirubin, indirect bilirubin, total protein, albumin, urea, creatinine. Additionally, routine blood indicators were evaluated, including haemoglobin, blood ketone bodies, white blood cell count, red blood cell count, and platelet count. Additionally, indicators of thyroid function are included, comprising free triiodothyronine, free thyroxine, thyrotropin, thyroid peroxidase antibodies, and thyroglobulin antibodies. Routine urine indicators are also provided, including pH, urine sugar, and urine ketone bodies.

(iii) Information on medication used during hospitalization: name of GLP-1AR drugs used, medication status (dosage, frequency, route, time and duration of administration), name of drugs used in combination, dosage, route of administration, course of treatment, and so on.

④Discharge examination data: basic information (weight, blood pressure, body temperature), glucose metabolism indicators (fasting blood glucose, postprandial 2h blood glucose, glycated hemoglobin), lipid metabolism indicators (triglycerides, total cholesterol, high-density lipoproteins, low-density lipoproteins), electrolyte indicators (potassium, sodium, magnesium, calcium ion concentration), indicators of hepatic and renal function (glutamic oxaloacetic aminase, glutamic oxaloacetic aminotransferase, total bile acid, total bilirubin, direct bilirubin, indirect bilirubin, total protein, albumin, urea, creatinine), routine blood indicators (hemoglobin, blood ketones, white blood cell count, red blood cell count, platelet count), and routine urinary indicators (pH, urinary glucose, urinary ketones).

(2) Collection of follow-up information

* Follow-up period and duration: follow-up of the included patients at the end of the 4th, 8th, 12th, and 16th weekends of drug administration, for a total of 12 weeks.

  * Format: telephone follow-up.

    ③ Follow-up information collection: Patient medication adherence: Morisky scale; Efficacy/safety: basic information, glucose metabolism indexes, lipid metabolism indexes, adverse drug reactions and other data from the beginning of drug administration to the end of the 4th, 8th, 12th and 16th weekends.

    (3) Recording and assessment of adverse drug reactions: The occurrence and severity of adverse drug reactions (ADRs) were recorded based on patients' active reports/chart descriptions and follow-up records, and the correlation between GLP-1RAs and adverse drug reactions was evaluated using the Noether Assessment Scale, and the severity was graded.

    (4) Study indicators Primary indicators: weight reduction from baseline, HbA1c Secondary indicators: medication adherence, change from baseline values of the four lipids, blood glucose fluctuation index, incidence of adverse drug reactions, total cost of GLP-1RAs during the follow-up cycle

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes;
* no study drug has been used in the last three months;
* Existing hypoglycemic programs include investigational drugs;
* Age ≥18 years old;
* The patient's demographic data, disease history, course records, laboratory test indicators, drug use and other information were complete;
* Sign informed consent.

Exclusion Criteria:

* persistent influenza, autoimmune disease, or other metabolic disease;
* There are obvious gastrointestinal diseases, gastrointestinal resection or malabsorption syndrome;
* diet drugs, glucocorticoids, drugs affecting gastrointestinal motility are being used;
* Patients with severe liver and kidney function impairment and patients with malignant tumors;
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type 2 diabetes
Sampling Method: Probability Sample
Enrollment: 492 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c compliance rate | 4, 8, 12, and 16 weeks after the start of medication
  HbA1c<7
Weight reduction from baseline | 4, 8, 12, and 16 weeks after the start of medication

CONTACTS AND LOCATIONS:
Overall Officials: Yining Dong, pharmacist, Principal Investigator — Shandong Third Hospital; Zhongming Wu, doctor, Principal Investigator — Endocrine and Metabolic Disease Hospital of Shandong First Medical University; Yue Liu, pharmacist, Principal Investigator — Shandong University of Traditional Chinese Medicine; Dandan Wu, pharmacist, Principal Investigator — Affiliated Hospital of Binzhou Medical College; Jing Peng, pharmacist, Principal Investigator — Jining Medical University; Qi Wang, pharmacist, Principal Investigator — Jinan Fifth People's Hospital; Zhaohui Meng, pharmacist, Principal Investigator — Jinan Laiwu People's Hospital; Dong wei Wang, doctor, Principal Investigator — Jinan Mental Health Center; Zhong Yuan, pharmacist, Principal Investigator — Jinan Municipal Hospital; Ming Xue, pharmacist, Principal Investigator — Jinan Hospital, Guang'anmen Hospital, China Academy of Traditional Chinese Medicine, China; Jing Lin, pharmacist, Principal Investigator — Shijhong District People's Hospital; Xingshan Wang, doctor, Principal Investigator — Changqing District Hospital of Traditional Chinese Medicine; Min Fan, pharmacist, Principal Investigator — Pingyin County People's Hospital; Xue Zheng, pharmacist, Principal Investigator — Zibo Center Hospital; Ming Xu, pharmacist, Principal Investigator — Zibo First Hospital; Yan Song, pharmacist, Principal Investigator — Zibo Municipal Hospital; Ruoxun Liu, pharmacist, Principal Investigator — Zibo Hospital of Traditional Chinese Medicine; Qing Zhao, doctor, Principal Investigator — Linzi District Maternal and Child Health Center; Zhenwei Chen, pharmacist, Principal Investigator — Yiyuan County People's Hospital; Zhiyan Li, pharmacist, Principal Investigator — Zaozhuang Municipal Hospital; Shenling Cheng, pharmacist, Principal Investigator — Tengzhou Central People's Hospital; Qixia Zhao, pharmacist, Principal Investigator — Zaozhuang Shanting District People's Hospital; Jintang Ning, pharmacist, Principal Investigator — Dongying People's Hospital; Juying Ding, pharmacist, Principal Investigator — Shengli Oilfield Hospital; Jiaxi Jiang, pharmacist, Principal Investigator — Haiyang People's Hospital; Guichun Wang, pharmacist, Principal Investigator — Longko People's Hospital; Zhentian Cheng, pharmacist, Principal Investigator — Weifang Yidu Center Hospital; Yueliang Ji, doctor, Principal Investigator — Fangzi District People's Hospital; Donglou Liang, pharmacist, Principal Investigator — Jining First People's Hospital; Li Zhang, pharmacist, Principal Investigator — QuFu People's Hospital; Guifeng Tan, doctor, Principal Investigator — Wenshang County People's Hospital; Ronghua Wang, pharmacist, Principal Investigator — Weihai Maternal and Child Health Center; Jianfang Liu, pharmacist, Principal Investigator — Rizhao People's Hospital; Xiangju Tian, doctor, Principal Investigator — Linyi Hospital of Traditional Chinese Medicine; Pengcheng Du, pharmacist, Principal Investigator — Shandong University Qilu Hospital, Dezhou Hospital; Fujian Xu, pharmacist, Principal Investigator — Heze Municipal Hospital; Deping Ho, pharmacist, Principal Investigator — Heze Third People's Hospital; Jingyong Xue, pharmacist, Principal Investigator — Heze Mudan People's Hospital; Lishun Yin, pharmacist, Principal Investigator — Heze Dingtao District People's Hospital; Shengmei Wei, pharmacist, Principal Investigator — Caoxian People's Hospital; Jing Meng, pharmacist, Principal Investigator — Shanxian Central Hospital; Ye Fan, pharmacist, Principal Investigator — Yuncheng County People's Hospital; Jingjing Zhang, pharmacist, Principal Investigator — Qingdao Eighth People's Hospital; Wenqian Han, pharmacist, Principal Investigator — Tai'an Central Hospital; Wenwen Lv, pharmacist, Principal Investigator — Affiliated Hospital of Binzhou Medical College; Tao Geng, pharmacist, Principal Investigator — The Second Affiliated Hospital of Shandong First Medical University; Fang Liu, pharmacist, Principal Investigator — Shengli Oilfield Hospital; Congrong Wang, pharmacist, Principal Investigator — Shandong Public Health Clinical Center; Ping Wang, pharmacist, Principal Investigator — Tengzhou Central People's Hospital; Yuxia Gao, pharmacist, Principal Investigator — Dongying Hospital Affiliated to Shandong University of Traditional Chinese Medicine (Dongying Hospital of Traditional Chinese Medicine); Bo Liu, pharmacist, Principal Investigator — Qingdao Central Hospital
Locations (1):
- Yan Li, Jinan, China

REFERENCES:
- [Result] Pratley RE, Aroda VR, Lingvay I, Ludemann J, Andreassen C, Navarria A, Viljoen A; SUSTAIN 7 investigators. Semaglutide versus dulaglutide once weekly in patients with type 2 diabetes (SUSTAIN 7): a randomised, open-label, phase 3b trial. Lancet Diabetes Endocrinol. 2018 Apr;6(4):275-286. doi: 10.1016/S2213-8587(18)30024-X. Epub 2018 Feb 1. PMID 29397376